CLINICAL TRIAL: NCT03148964
Title: Multicentric Cohort of HIV-1 (Human Immunodeficiency Virus 1) Primary Infection Cohort ANRS CO6 PRIMO
Brief Title: Primary Infection Cohort
Acronym: PRIMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS CO6 PRIMO
Record Dates: First submitted 2017-04-12; First posted 2017-05-11 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, full blood, serum, lymphocytes and cells samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow-up Arm: Blood sampling only
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — Blood Sampling at J0, M1, M3, M6, M12, M24 and every 12 months until the end of the study

SUMMARY:
Open, prospective, multicenter French cohort study enrolling subjects aged of 15 years or more, during or immediately after HIV-1 primary infection. This cohort was organized from the outset to be highly multidisciplinary, bringing together immunologists, virologists, clinicians and epidemiologists.

DETAILED DESCRIPTION:
Objectives: Follow up of patients infected by HIV-1 for less than three months.

1. Improve the physiological and pathological knowledge of primary HIV infection

   * Study of the immune mechanisms involved early after infection
   * Kinetics of viral replication and establishment of cellular reservoirs at an early stage
   * Relationships between virological markers and immune response kinetics
   * Impact of resistance mutations, subtype and tropism on the disease progression and the response to treatment
   * Study of sub-groups of specific patients followed since primary infection, spontaneous or post treatment controllers, subjects with specific HLA
2. Assessing the impact of early, transient or prolonged treatment versus deferred treatment on the long-term prognosis of patients followed since primary infection, in terms of activation / inflammation and decrease in viral reservoirs
3. Contribute to knowledge in the epidemiology of HIV infection:

   * Modes of transmission
   * Sexual behavior after HIV diagnosis
   * Calendar trend of transmitted viral strains diversity (ARV resistance and subtypes)
   * Calendar trend of marker levels measured at primary infection
4. Contribute to national recommendations for therapeutic care, evaluate their implementation
5. Use observational data from the cohort for the development of therapeutic clinical trials at primary infection

ELIGIBILITY:
Inclusion Criteria:

* symptomatic or asymptomatic HIV-1 primary infection.
* Infection date based on one of the following criteria:

  1. Positive p24 antigenemia or detectable plasma HIV RNA with a negative ELISA within the previous six weeks.
  2. Positive p24 antigenemia or detectable plasma HIV RNA with a positive ELISA and negative Western Blot within the previous six weeks.
  3. Positive p24 antigenemia or detectable plasma HIV RNA or positive ELISA with incompleted Western Blot (no anti-p34 and/or anti-p68) within the previous six weeks.
  4. Positive ELISA with a negative ELISA within the last three months.
* Age≥ 15 years old at the enrollment.
* Naive of antiretroviral treatment except for transient treatment taken in the context of PMTCT, Pre-exposition prophylaxis or Post Exposition Prophylaxis.
* Affiliate or beneficiary of a social security system (State Medical Assistance is not a social security scheme).

Exclusion Criteria:

* Inability to give informed consent.
* Predictable difficult follow-up.
* Contraindication to repeated blood samples.
* Under protection (saving) of justice
* Life-threatening pathology (deferred inclusion is possible)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-1 infected patients
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 1996-10 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Improve the physiological, pathological and virological knowledge of primary HIV infection | up to 25 years
  * Study of the immune mechanisms involved early after infection
  * Kinetics of viral replication and establishment of cellular reservoirs at an early stage
  * Relationships between virological markers and immune response kinetics
  * Impact of resistance mutations, subtype and tropism on the disease progression and the response to treatment
  * Study of sub-groups of specific patients followed since primary infection, spontaneous or post treatment controllers, subjects with specific HLA

SECONDARY OUTCOMES:
The impact of early, transient or prolonged treatment versus deferred treatment on the long-term prognosis of patients followed since primary infection, in terms of activation / inflammation | up to 25 years
Contribute to knowledge in the epidemiology of HIV infection | up to 25 years
  * Modes of transmission
  * Sexual behavior after HIV diagnosis
  * Calendar trend of transmitted viral strains diversity (ARV resistance and subtypes)
  * Calendar trend of marker levels measured at primary infection
Contribute to national recommendations for therapeutic care and evaluate their implementation | up to 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Meyer, Professor, Principal Investigator — CESP-INSERM U1018
Locations (1):
- Laurence Meyer, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baltes V, de Boissieu P, Champenois K, Luan L, Seng R, Essat A, Novelli S, Spire B, Molina JM, Goujard C, Meyer L; ANRS PRIMO cohort study group. Sexual behaviour and STIs among MSM living with HIV in the PrEP era: the French ANRS PRIMO cohort study. J Int AIDS Soc. 2024 Mar;27(3):e26226. doi: 10.1002/jia2.26226. PMID 38462760